CLINICAL TRIAL: NCT06978114
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1+PD-1/PD-L1 Monoclonal Antibody in Patients With Advanced Biliary Tract Cancer
Brief Title: A Study of BL-B01D1+PD-1/PD-L1 Monoclonal Antibody in Patients With Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-10
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1+Pembrolizumab (Experimental): Participants receive BL-B01D1+Pembrolizumab in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: Pembrolizumab — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a clinical study to explore the efficacy and safety of BL-B01D1+PD-1/PD-L1 monoclonal antibody in patients with advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Patients with advanced biliary tract cancer confirmed by histology or cytology;
6. Patients must provide a documented tumor tissue specimen of the primary or metastatic tumor within 3 years for PD-L1 testing and other testing;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG score 0-1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. Organ function level must meet the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Patients with active central nervous system metastases;
2. Who had participated in any other clinical trial within 4 weeks before the trial dose;
3. Received anti-tumor therapy such as chemotherapy, radiotherapy and biological therapy within 4 weeks before the first use of study drug;
4. Had undergone major surgery (investigator-defined) within 4 weeks before the first dose;
5. Had received immunotherapy and developed grade ≥3 irAE or grade ≥2 immune-related myocarditis;
6. Use of immunomodulatory drugs within 14 days before the first dose of study drug;
7. Systemic corticosteroids or immunosuppressive agents were required within 2 weeks before the study administration;
8. Pulmonary disease grade ≥3 according to NCI-CTCAE v5.0; A history of ILD/pulmonary inflammation requiring steroid treatment;
9. Severe systemic infection occurred within 4 weeks before screening;
10. Patients at risk for active autoimmune disease or with a history of autoimmune disease;
11. Other malignant tumors within 5 years before the first dose;
12. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
13. Poorly controlled hypertension by two antihypertensive drugs with different mechanisms;
14. Diabetic patients with poor glycemic control;
15. Had a history of severe cardiovascular and cerebrovascular diseases;
16. Previous history of autologous or allogeneic stem cell, bone marrow or organ transplantation;
17. Subjects with clinically significant bleeding or significant bleeding tendency within the preceding 4 weeks were screened;
18. Patients with massive or symptomatic effusions or poorly controlled effusions;
19. Imaging examination showed that the tumor had invaded or wrapped around the chest, neck, pharynx and other large arteries or invaded the pericardium and heart;
20. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
21. Prior treatment with an ADC drug with a topoisomerase I inhibitor as a toxin;
22. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of the trial drug;
23. The cumulative dose of anthracyclines > 360 mg/m2 in previous (new) adjuvant therapy;
24. Pregnant or lactating women;
25. Who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
26. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China